CLINICAL TRIAL: NCT04134637
Title: The Analgesic Effect of Ultrasound Guided Bilateral Pecto Intercostal Fascial Plane Block on Sternal Wound Pain After Open Heart Surgeries
Brief Title: Bilateral Pecto Intercostal Fascial Plane Block After Open Heart Surgeries
Acronym: PIFB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, lecturer of anesthesia and intensive care, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: D178
Record Dates: First submitted 2019-07-12; First posted 2019-10-22 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Pain, Chest
Keywords: pecto intercostal fascial plane block; sternotomy
MeSH Terms: conditions — Chest Pain | interventions — Ultrasonography; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIFB group (Experimental): For carrying out PIFB bilaterally the skin on either side of the sternum will be prepared with povidone iodine solution. Then a linear ultrasound probe will be placed on the right and left sides at 2 cm from the sternal body.
  A 22 gauge, 4 inch needle will be advanced until contacting the 4th costal cartilage following the lower edge of US probe, directing the tip from the bottom of the sternum and positioning the needle tip between the pectoralis major and the external intercostal muscles. Group A will receive twenty milliliters of a solution of 0.25% bupivacaine plus epinephrine (5 mcg/ml). Boluses of 5 ml are introduced to perform hydrodissection of the interfascial plane.
  Interventions: Device: ultrasound; Drug: Bupivacaine Hydrochloride 5 MG/ML
- control group (No Intervention): the block will not be given

INTERVENTIONS:
Device: ultrasound — in the PIFB group linear ultrasound (Philips clear vue350,Philips healthcare,Andover MAO1810,USA,Machine Identification number:1385,Nile medical center,service@nilemed.net) probe will be used.
  Arms: PIFB group
Drug: Bupivacaine Hydrochloride 5 MG/ML — twenty milliliters of a solution of 0.25% bupivacaine in the PIFB group
  Other Names: sunnypivacaine
  Arms: PIFB group

SUMMARY:
The objective is to test the effect of pecto intercostal fascial plane block (PIFB) as regard its impact on pain after sternotomy involved open heart surgery. The authors hypothesize that bilateral PIFB can reduce pain resulting from sternotomy following open heart surgeries.

DETAILED DESCRIPTION:
Pain following cardiac surgery is caused by many factors; sternotomy, chest wall retraction, opening of the pericardium, internal mammarian artery harvesting, saphenous vein harvesting, surgical manipulation of the parietal pleura, chest tube insertion and other musculoskeletal trauma occurring during surgery.

The pain following cardiac surgery is mainly attributed to sternotomy, with its peak during the first two days after the operation. Poststernotomy pain is not well tolerated by patients and may be accompanied by adverse postoperative events including delirium, hypertension, tachycardia, arrhythmia, respiratory complications, and persistent postsurgical pain.

Commonly pain management after cardiac surgery has been achieved using opiate analgesics. However, opiates have some dose-related side-effects such as nausea, constipation, vomiting, dizziness, mental confusion and respiratory depression, which may influence patient recovery and may delay discharge after surgery.

The pecto-intercostal fascial block (PIFB) was recently introduced by de la Torre et al for anesthesia during breast surgery. Local anesthetic is infiltrated into the interfascial plane separating pectoralis major and the intercostal muscles lateral to the sternum to anesthetize the anterior cutaneous branches of the intercostal nerves.

The pecto-intercostal fascial plane block can cover anterior branches of the intercostal nerves from the 2nd to 6th dermatomes with a single injection bilaterally, same as the transversus thoracic muscle plane block .

anesthetic management: All patients will be preoperatively examined and investigated by complete blood count, coagulation profile, renal and kidney functions and electrolytes. Electrocardiography, chest x ray and echocardiography will be routinely done. Coronary angiography and carotid arterial duplex will be requested in patients prepared for CABG.

Patient will be premedicated by intramuscular injection of 10mg morphine in the morning of the operation. Before induction of anesthesia, a five-lead electrocardiography system will be applied to monitor heart rate, rhythm, and ST segments (leads II and V5). A pulse oximeter probe will be attached, and a peripheral venous cannula will be placed. For measurement of arterial pressure and blood sampling, a 20 G cannula will be inserted into either right or left radial artery under local anesthesia. General anesthesia will be induced by midazolam 2-5 mg, fentanyl (10 μg/kg), propofol (3-4mg/Kg), followed by atracurium (0.5 mg/kg).

Trachea will be intubated, patients will be mechanically ventilated with oxygen in air so as to achieve normocarbia. This will be confirmed by radial arterial blood gas analysis. An esophageal temperature probe and a Foley catheter will also be placed.

For drug infusion, a triple-lumen central venous catheter will be inserted via the right internal jugular vein.

Anesthesia will be maintained by inhaled Isoflurane 0.4 to 1% and atracurium infusion at a rate of 0.5 mg/kg/h for continued muscle relaxation. During extracorporeal circulation, patients will receive propofol infusion at a rate of 100-200 mg/h in addition to atracurium infusion.

Before initiation of cardiopulmonary bypass (CPB), the patients will receive intravenously tranexamic acid (2 g) and heparin (300-500 units/kg body weight) to achieve an activated clotting time > 480 s. CPB will be instituted via an ascending aortic cannula and a two-stage right atrial cannula. Before, during, and after CPB (pump blood flow: 2.4 l/min/m2), mean arterial pressure will be adjusted to exceed 60 mmHg. Cardiac arrest will be induced with cold antegrade blood cardioplegia or warm intermittent antegrade crystalloid cardioplegia. Lactate-enriched Ringer's solution will be added to the CPB circuit to maintain reservoir volume when needed, and packed red blood cells will be added when hemoglobin concentration decrease to less than 7 g/dl.

After rewarming the patient to 37°C and separation from CPB, reversal of heparin by protamine sulfate (1:1), and sternal closure will be achieved.

All patients then will be shifted to the intensive care unit (ICU) after the surgery and managed with the institution's ICU protocol for postoperative pain management and ventilation. The postoperative analgesia protocol involves the use of intravenous morphine or morphine equivalent dose of 5to 10 mg/kg bolus as required. Criteria for administration will be signs of sympathetic stimulation in the form of undue tachycardia, a rise in mean arterial pressure (rise of >20% from the baseline).

Tracheal extubation will be performed when the patient met the following criteria: awake/arousable, hemodynamically stable, no active bleeding, warm peripheries, and satisfactory arterial blood gas with an FiO2 < 0.5,pressure support on ventilator reduced to 10 Cm H2O,Positive End Expiratory Pressure 5-7 CmH2O, no electrolyte abnormalities, minimal inotropic support, or no escalation in inotropic support.

Statistical analysis Sample size was calculated using (G power version 3). Minimal sample size of patients was 31 in each group needed to get power level 0.90, alpha level 0.05 and 30% as a difference between the two groups in the morphine consumption after the intervention. To overcome problem of loss of follow up, calculated sample size was increased by 10% to reach 35 in each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective cardiovascular surgery for coronary artery bypass grafting or valve replacement involving median sternotomy

Exclusion Criteria:

* Patients with emergency surgeries.
* Allergy to drug used.
* Patients with prolonged Cardio-Pulmonary Bypass time (>120 min).
* Preoperative poor left ventricular function (ejection fraction <40%).
* Body Mass Index >40.
* Systemic infections or infections at site of injection.
* Prolonged ICU stay over 24 hours for different reasons i.e.re-do surgery, heart failure etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Cumulative morphine consumption | 24 hours postoperative
  in milligram

SECONDARY OUTCOMES:
postoperative sternal wound pain degree | 4 hours after extubation
  Objective pain score (1:pain at rest , 2:Pain free at rest, 3:Pain free when deep breathing, but pain when coughing, 4:Pain free, even when coughing
  1 (worst) to 4 (best) not summed
postoperative sternal wound pain degree | 8 hours after extubation
  Objective pain score (1:pain at rest , 2:Pain free at rest, 3:Pain free when deep breathing, but pain when coughing, 4:Pain free, even when coughing
  1 (worst) to 4 (best) not summed
postoperative sternal wound pain degree | 12 hours after extubation
  Objective pain score (1:pain at rest , 2:Pain free at rest, 3:Pain free when deep breathing, but pain when coughing, 4:Pain free, even when coughing
  1 (worst) to 4 (best) not summed
postoperative sternal wound pain degree | 16 hours after extubation
  Objective pain score (1:pain at rest , 2:Pain free at rest, 3:Pain free when deep breathing, but pain when coughing, 4:Pain free, even when coughing
  1 (worst) to 4 (best) not summed
postoperative sternal wound pain degree | 20 hours after extubation
  Objective pain score (1:pain at rest , 2:Pain free at rest, 3:Pain free when deep breathing, but pain when coughing, 4:Pain free, even when coughing
  1 (worst) to 4 (best) not summed
postoperative sternal wound pain degree | 24 hours after extubation
  Objective pain score (1:pain at rest , 2:Pain free at rest, 3:Pain free when deep breathing, but pain when coughing, 4:Pain free, even when coughing
  1 (worst) to 4 (best) not summed
Heart rate | 1 minute before induction of anesthesia, 5 minutes after induction of anesthesia then every 30 minutes for 8 times
  in beat per minute
systolic blood pressure | 1 minute before induction of anesthesia, 5 minutes after induction of anesthesia then every 30 minutes for 8 times
  in millimeter mercury
diastolic blood pressure | 1 minute before induction of anesthesia, 5 minutes after induction of anesthesia then every 30 minutes for 8 times
  in millimeter mercury
peripheral oxygen saturation | 1 minute before induction of anesthesia, 5 minutes after induction of anesthesia then every 30 minutes for 8 times
  in percentage by pulse oximetry
heart rate | 1 minute after admission in ICU then every 4 hours for 6 times then every 8 hours for 3 times
  in beat per minute
systolic blood pressure | 1 minute after admission in ICU then every 4 hours for 6 times then every 8 hours for 3 times
  in millimeter mercury
diastolic blood pressure | 1 minute after admission in ICU then every 4 hours for 6 times then every 8 hours for 3 times
  in millimeter mercury
peripheral oxygen saturation | 1 minute after admission in ICU then every 4 hours for 6 times then every 8 hours for 3 times
  in percentage by pulse oximetry
incidence of Myocardial infarction | 1 minute after ICU admission
  number
incidence of postoperative pericardial effusion | 1 minute after ICU admission
  number
incidence of heart failure requiring inotropic support | 1 minute after ICU admission
  number
incidence of atrial fibrillation | 1 minute after ICU admission
  number
partial pressure of oxygen | 1 minute after insertion of arterial cannula
  by mmhg in arterial blood gases
partial pressure of oxygen | 1 minute after extubation
  by mmhg in arterial blood gases
partial pressure of oxygen | 6 hour after extubation
  by mmhg in arterial blood gases
partial pressure of oxygen | 12 hour after extubation
  by mmhg in arterial blood gases
incidence of cerebral stroke | 1 minute after ICU admission up to 2 days
  number
incidence of cerebral bleeding | 1 minute after ICU admission up to 2 days
  number
Gastrointestinal bleeding | 1 minute after ICU admission up to 2 days
  number
blood component requirements | 1 minute after ICU admission up to 2 days
  number
incidence of sternal complications. | 1 minute after ICU admission up to 2 days
  number
hospital stay | 1 minute after ICU admission up to 2 days
  in days

OTHER OUTCOMES:
Age | 2 hours before operation
  in years
body mass index | 2 hours before operation
  kilogram/square meter

CONTACTS AND LOCATIONS:
Overall Officials: Maged L Boules, MD, Study Chair — Faculty of medicine, Fayoum university; Mohamed A Hamed, MD, Study Director — Faculty of medicine, Fayoum university
Locations (1):
- Fayoum university hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang AP, Sakata RK. [Pain after sternotomy - review]. Rev Bras Anestesiol. 2016 Jul-Aug;66(4):395-401. doi: 10.1016/j.bjan.2014.09.003. Epub 2015 Mar 18. Portuguese. PMID 25796483
- [Background] Mazzeffi M, Khelemsky Y. Poststernotomy pain: a clinical review. J Cardiothorac Vasc Anesth. 2011 Dec;25(6):1163-78. doi: 10.1053/j.jvca.2011.08.001. Epub 2011 Sep 29. No abstract available. PMID 21955825
- [Background] Chandrakantan A, Glass PS. Multimodal therapies for postoperative nausea and vomiting, and pain. Br J Anaesth. 2011 Dec;107 Suppl 1:i27-40. doi: 10.1093/bja/aer358. PMID 22156268
- [Background] Del Buono R, Costa F, Agro FE. Parasternal, Pecto-intercostal, Pecs, and Transverse Thoracic Muscle Plane Blocks: A Rose by Any Other Name Would Smell as Sweet. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):791-792. doi: 10.1097/AAP.0000000000000464. No abstract available. PMID 27776103
- [Background] Ohgoshi Y, Ino K, Matsukawa M. Ultrasound-guided parasternal intercostal nerve block. J Anesth. 2016 Oct;30(5):916. doi: 10.1007/s00540-016-2202-5. Epub 2016 Jun 20. No abstract available. PMID 27325411